CLINICAL TRIAL: NCT00293839
Title: Comparison of the Efficacy and Tolerability of DITROPAN XL and DETROL LA in the Treatment of Overactive Bladder
Brief Title: Efficacy and Tolerability of DITROPAN XL (Oxybutynin Chloride) Versus DETROL LA (Tolterodine Tartrate) in Treatment of Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004570
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Urinary Incontinence
Keywords: bladder; overactive
MeSH Terms: conditions — Urinary Incontinence | interventions — oxybutynin

INTERVENTIONS:
Drug: oxybutynin chloride

SUMMARY:
The purpose of this study is to compare the efficacy of DITROPANÂ® XL (oxybutynin chloride) Extended-Release Tablets and DETROLÂ® LA (tolterodine tartrate extended-release capsules) in the reduction of urge urinary incontinence episodes during a 12-week treatment period in patients with overactive bladder. The secondary objective is to compare the tolerability of DITROPANÂ® XL (oxybutynin chloride) and DETROLÂ® LA (tolterodine tartrate) during a 12-week treatment period.

DETAILED DESCRIPTION:
The objective of this study is to compare the efficacy and tolerability of DITROPAN® XL 10 mg once-daily and DETROL® LA 4 mg once-daily in the reduction of urge urinary incontinence episodes in female patients with overactive bladder. This is a multicenter, randomized, double-blind, parallel-group study with two active treatments. Screened patients are qualified for the study based on information obtained from seven consecutive 24-hour urinary diaries completed during the Baseline Week, and other eligibility criteria. Qualifying patients receive 12 weeks of treatment with DITROPAN® XL or DETROL® LA, with clinical visits at the end of Weeks 2, 4, 8, and 12.

Safety evaluations during the study include the collection of adverse events, laboratory tests including blood chemistry and urinalysis, physical examinations, vital signs (blood pressure and heart rate) and post-void residual urine volume. Over-encapsulated DITROPAN® XL, 10 mg tablets once-daily by mouth or over-encapsulated DETROL® LA, 4 mg capsules once daily by mouth. The treatment phase of the study runs for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are able to differentiate urinary incontinence episodes associated with urgency from urinary incontinence episodes not associated with urgency
* during the 7 day baseline period have 21 to 60 urge urinary incontinence (Urge-UI) episodes, a greater number of Urge-UI episodes than urinary incontinence not associated with urge, and an average of 10 or more voids per 24 hours
* are in good general health as determined by medical history, physical examination (general, genital, pelvic, and rectal), laboratory tests and urinalysis
* if taking antihypertension medication, must be on a stable dose
* and if of child-bearing potential, practicing an acceptable method of birth control, and must have a negative pregnancy test at Visit 2 and Visit 3

Exclusion Criteria:

* Participants with known, treatable genitourinary conditions (identified on history or on examination) that may cause incontinence (e.g., urinary tract infection, interstitial cystitis, urinary tract obstruction, urethral diverticulum, bladder tumor, bladder stone)
* have given birth or have had pelvic, vaginal or bladder surgery less than 6 months before study enrollment
* with a second post-void residual urine volume > 150 mL at the time of screening (determined by abdominal ultrasound)
* with significant medical problems or other organ abnormality that places them at risk from participating in the study or at a significant risk of developing complete urinary retention
* with significant impairment of the liver or kidneys as determined by laboratory assessments or hematuria (red blood cells in microscopic urinalysis)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
The number of weekly urge urinary incontinence (Urge-UI) episodes at week 12, adjusted for the baseline value

SECONDARY OUTCOMES:
The number of total urinary incontinence (Total-UI) episodes at week 12; Void frequency at week 12; Urge-UI ,Total-UI, and Void frequence at weeks 2, 4, and 8; tolerability of the treatments during the 12-week treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Result] Diokno AC, Appell RA, Sand PK, Dmochowski RR, Gburek BM, Klimberg IW, Kell SH; OPERA Study Group. Prospective, randomized, double-blind study of the efficacy and tolerability of the extended-release formulations of oxybutynin and tolterodine for overactive bladder: results of the OPERA trial. Mayo Clin Proc. 2003 Jun;78(6):687-95. doi: 10.4065/78.6.687. PMID 12934777